CLINICAL TRIAL: NCT06649175
Title: Effect of Kinetic Chain Exercises on Muscle Strength, Joint Position Sense and Quality of Life in Children with Haemophilia.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmein Nabil Mohamed El Tanany, Physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005128
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-03

CONDITIONS: Hemophilia a; Muscle Strength; Joint Position Sense; Quality of Life (QOL)
MeSH Terms: conditions — Hemophilia A | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group(A):exercise group. (Active Comparator): Control Group (A): will receive the traditional physical therapy (PT) program for one hour two times weekly for six successive weeks.
  Intervention: traditional physical therapy program.
  Interventions: Other: Exercise
- Group(B): modified exercise group. (Active Comparator): Group (B): will receive a program of close kinetic chain exercises for 30 min.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Close kinetic chain (CKC) exercises :
  1. Supine wall push exercise: Start position: supine with the both leg against wall, other limb straight. Exercise action: push against wall for thirty seconds.
  2. Wall push against Swiss ball exercise: Start position: Supine with a Swiss ball between patient's legs and the wall. Exercise action: push against the wall for thirty seconds.
  3. Supine half bridging exercise: Start position: Lying on back, knees bent Exercise action: keeping spine neutral and hinging up from the hips, move into a bridge.
  Other Names: Close Kinetic Chain Exercise (CKC)
  Arms: Group(B): modified exercise group.
Other: Exercise — Control Group (A): will receive the traditional physical therapy (PT) , the traditional physical therapy program will include the following:
  * Stretching exercise for shortening muscle of lower limbs (LL) mainly (hip flexors, adductors, knee flexors and ankle planter flexors).
  * Balance training from standing while giving perturbations.
  * Balance board training.
  * Step ups: repeated stepping anteriorly and laterally onto a step with both legs alternatively, progressing to higher step and decreasing upper extremity support.
  * Forward and backward walking (with or without handheld mobility devices).
  * Side walking (with or without handheld mobility devices).
  * Walking in astride line (with or without handheld mobility devices).
  Other Names: Traditional physical therapy program
  Arms: group(A):exercise group.

SUMMARY:
The goal of this clinical trial is to learn if there are effect of close kinetic chain exercises on muscle strength, joint position sense and Quality of life in children with haemophilia? Null hypothesis

It will be hypothesized that:

There is no effect of close kinetic chain exercises on muscle strength, joint position sense and Quality of life in children with haemophilia.

DETAILED DESCRIPTION:
Sample size estimation will be carried out to determine the recruited number of children selected randomly from Out Patient clinic of Atfal Misr hospital, Cairo governorate to participate in this study. The study targets male children with hemophilia A.

They will be selected based on the following:

Inclusion criteria:

1. Their chronological age will be 5-7yeasr.
2. All children will receive prophylaxis therapy.
3. They will able to stand and walk independently.
4. They will be able to follow instructions during evaluation and treatment.

Exclusive criteria:

The children will be excluded if they have one of the following:

1. Visual or auditory problem.
2. Radiographic changes as bone erosions, destruction, or joint subluxation, or congenital or acquired skeletal deformities in both lower limbs.
3. Surgical procedures performed six weeks prior to or during study.
4. Bleeding in joint 2 week prior to assessment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Their chronological age will be 5-7yeasr. 2. All children will receive prophylaxis therapy. 3. They will able to stand and walk independently. 4. They will be able to follow instructions during evaluation and treatment.

Exclusion Criteria:

* The children will be excluded if they have one of the following:

  1. Visual or auditory problem.
  2. Radiographic changes as bone erosions, destruction, or joint subluxation, or congenital or acquired skeletal deformities in both lower limbs.
  3. Surgical procedures performed six weeks prior to or during study.
  4. Bleeding in joint 2 week prior to assessment.

Ages: 5 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
a) Assessment of muscle strength: | baseline only
  The isometric muscle strength of bilateral knee extensors muscles will be measured with a handheld dynamometer.

SECONDARY OUTCOMES:
b) Assessment of knee joint position sense. | baseline only
  Knee joint position sense will be measures with a Saunders digital inclinometer.

OTHER OUTCOMES:
c) Assessment of Quality of life. | baseline only
  The Haemo-QoL questionnaire is a quality of life assessment instrument for children with haemophilia.

CONTACTS AND LOCATIONS:
Locations (1):
- Out Patient clinic of Atfal Misr hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided